CLINICAL TRIAL: NCT00759824
Title: A Phase II Study of Doxorubicin, Cyclophosphamide and Vindesine With Valproic Acid in Patients With Refractory or Relapsing Small Cell Lung Cancer After Platinum Derivatives and Etoposide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01081
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Small cell lung carcinoma; Valproic acid; Adriamycin; Cyclophosphamide; Vindesine; Second-line chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Doxorubicin; Cyclophosphamide; Vindesine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Chemotherapy regimen (adriamycin, cyclophosphamide, vindesine) plus valproic acid
  Interventions: Drug: Adriamycin, cyclophosphamide, vindesine, valproic acid

INTERVENTIONS:
Drug: Adriamycin, cyclophosphamide, vindesine, valproic acid — Adriamycin 45 mg/m² day 1 IV Cyclophosphamide 1 g/m² day 1 IV Vindesine 3 mg/m² day 1 IV Valproic acid 20-30 mg/kg/day from day -7 until the end of treatment, orally

SUMMARY:
The primary aim of this study is to determine if the addition of valproic acid to a combination of adriamycin, cyclophosphamide and vindesine could increase progression-free survival in patients relapsing after first-line chemotherapy including platinum derivatives, cisplatin or carboplatin, and etoposide.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of small-cell lung cancer (SCLC)
* SCLC refractory to prior chemotherapy regimen including platinum derivatives (cisplatin or carboplatin) and etoposide, either primary refractory (immediate progression or recurrence less than 3 months after the end of previous chemotherapy) or secondary refractory (sensitive patients to platinum plus etoposide in first-line, progressing or recurring less than 3 months after reintroduction of the same chemotherapy).
* At least one evaluable or measurable lesion
* Availability for participating in the detailed follow-up of the protocol
* Signed informed consent.

Exclusion Criteria:

* Patient who were previously treated with anthracyclin or vinca-alcaloid derivatives or cyclophosphamide
* Performance status < 60 on the Karnofsky scale
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or of the bladder or cured malignant tumour (more than 5-year disease free interval)
* A history of prior HIV infection
* Polynuclear cells < 2,000/mm³
* Platelet cells < 100,000/mm³
* Abnormal coagulation tests (aPTT, PTT, prothrombin time) and/or decreased fibrinogen
* Serum bilirubin >1.5 mg/100 ml
* Transaminases more than twice the normal range
* Serum creatinine > 1.5 mg/100 ml
* Recent myocardial infarction (less than 3 months prior to date of diagnosis)
* Congestive cardiac failure (ejection fraction of the left ventricle < 50%) or uncontrolled cardiac arrhythmia
* Uncontrolled infectious disease
* Active epilepsy needing a specific treatment
* Concomitant treatment with IMAO, carbamazepine, mefloquine, phenobarbital, primidone, phenytoïn, lamotrigine, zidovudine
* Pregnancy or refusal to use active contraception
* A known allergy to valproic acid and/or doxorubicin, cyclophosphamide, vindesine
* Serious medical or psychological factors which may prevent adherence to the treatment schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Six-months progression-free survival | The period between the day of registration and the date of first progression

SECONDARY OUTCOMES:
Survival | Survival will be dated from the date of registration
Response rate | Every three cycles of chemotherapy
Toxicity | After each course of chemotherapy and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, Study Chair — European Lung Cancer Working Party
Locations (5):
- Belgium (5):
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Department of Pneumology Centre Hospitalier de Mouscron, Mouscron

REFERENCES:
- See also: (Click here for more information on the protocol) — http://www.elcwp.org